CLINICAL TRIAL: NCT07130006
Title: Preoperative Use of Peripheral Nerve Blocks in Elderly Patients With Hip Fractures: a Factorial Randomized Clinical Trial
Brief Title: Preoperative Use of Peripheral Nerve Blocks in Elderly Patients With Hip Fractures
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital of Split (Other)
Responsible Party: Principal Investigator, Ana Saric Jadrijev, MD, Anaesthesiology, Reanimatology and Intensive Medicine Specialist, Principal Investigator, University Hospital of Split
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2181-147/01-06/LJ.Z.-25.02.
Record Dates: First submitted 2025-06-22; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Fractures, Hip; Femoral Neck Fractures; Intertrochanteric Fractures; Subtrochanteric Fractures; Aged; Frail Older Adults; Elderly
Keywords: elderly; ultrasound-guided; peripheral nerve blocks; intravenous fentanyl; spinal anaesthesia; EQ-5D-5L; visual analog scale; pain at rest; dynamic pain; hip fracture surgery
MeSH Terms: conditions — Hip Fractures; Femoral Neck Fractures | interventions — Anesthesia, Spinal; Fentanyl

STUDY DESIGN:
Intervention Model Description: Factorial randomized controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Respondents will not know to which group they have been randomized, nor will the surgeons, anesthesiology residents, nor nurses on the ward. Anesthesiologists will be familiar with all the items and will therefore be considered as the study supervisors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Intracapsular hip fracture FEMORAL BLOCK (Active Comparator): Patients with intracapsular hip fracture. The fracture pattern is verified with a native X-ray image of the broken hip in 2 projections. Peripheral nerve block and spinal anesthesia are administered for partial endoprothesis of hip fracture.
  Interventions: Procedure: FN and LFCN peripheral nerve blocks with spinal anesthesia
- Intracapsular hip fracture PENG BLOCK (Active Comparator): Patients with intracapsular hip fracture. The fracture pattern is verified with a native X-ray image of the broken hip in 2 projections. Peripheral nerve block and spinal anesthesia are administered for partial endoprothesis of hip fracture.
  Interventions: Procedure: PENG and LFCN peripheral nerve blocks with spinal anesthesia
- Intracapsular hip fracture FASCIA ILIACA BLOCK (Active Comparator): Patients with intracapsular hip fracture. The fracture pattern is verified with a native X-ray image of the broken hip in 2 projections. Peripheral nerve block and spinal anesthesia are administered for partial endoprothesis of hip fracture.
  Interventions: Procedure: FIC peripheral nerve block with spinal anesthesia
- Intracapsular hip fracture FENTANYL (Active Comparator): Patients with intracapsular hip fracture. The fracture pattern is verified with a native X-ray image of the broken hip in 2 projections. Fentanyl intravenously and spinal anesthesia are administered for partial endoprothesis of hip fracture.
  Interventions: Procedure: Fentanyl (IV) with spinal anesthesia
- Extracapsular hip fracture FEMORAL BLOCK (Active Comparator): Patients with extracapsular hip fracture. The fracture pattern is verified with a native X-ray image of the broken hip in 2 projections. Peripheral nerve blocks and spinal anesthesia are administered for osteosinthesis of hip fracture.
  Interventions: Procedure: FN and LFCN peripheral nerve blocks with spinal anesthesia
- Extracapsular hip fracture PENG BLOCK (Active Comparator): Patients with extracapsular hip fracture. The fracture pattern is verified with a native X-ray image of the broken hip in 2 projections. Peripheral nerve blocks and spinal anesthesia are administered for osteosinthesis of hip fracture.
  Interventions: Procedure: PENG and LFCN peripheral nerve blocks with spinal anesthesia
- Extracapsular hip fracture FASCIA ILIACA BLOCK (Active Comparator): Patients with extracapsular hip fracture. The fracture pattern is verified with a native X-ray image of the broken hip in 2 projections. Peripheral nerve block and spinal anesthesia are administered for osteosinthesis of hip fracture.
  Interventions: Procedure: FIC peripheral nerve block with spinal anesthesia
- Extracapsular hip fracture FENTANYL (Active Comparator): Patients with extracapsular hip fracture. The fracture pattern is verified with a native X-ray image of the broken hip in 2 projections. Fentanyl intravenously and spinal anesthesia are administered for osteosinthesis of hip fracture.
  Interventions: Procedure: Fentanyl (IV) with spinal anesthesia

INTERVENTIONS:
Procedure: PENG and LFCN peripheral nerve blocks with spinal anesthesia — At first, one needs to detect hyperechogenic iliopsoas notch and psoas tendon, between anterior inferior iliac spine and iliopubic eminence. Then needle needs to be inserted in-plane and 20mL of levobupivacaine 0.25% administered along the fascial plane. Additionally, after identification of sartorius muscle, 5mL of levobupivacaine 0.5% need to be administered in a space between sartorius and tensor fascia latae muscles where lateral femoral cutaneous nerve can be identified as a hyperechoic structure. Single shot needle, with bevel up, will be visible all the time, in plane technique will be used. The spread of the local anesthetic will appear hypoechoic on ultrasound. Curvilinear probe will be used.
  For spinal anesthesia levobupivacaine will be placed in the subarachnoid space at lumbar vertebrae 3/4 level using 25 G spinal needle.
  Arms: Extracapsular hip fracture PENG BLOCK; Intracapsular hip fracture PENG BLOCK
Procedure: FN and LFCN peripheral nerve blocks with spinal anesthesia — At first, one needs to detect both femoral artery and vein medial to it. Then needle needs to be inserted in-plane and 15mL of levobupivacaine 0.5% need to be administered underneath fascia iliaca, lateral to femoral nerve. Additionally, after identification of sartorius muscle, 5mL of levobupivacaine 0.5% need to be administered in a space between sartorius and tensor fascia latae muscles, where lateral femoral cutaneous nerve can be identified as a hyperechoic structure. Single shot needle, with bevel up, will be visible all the time, in plane technique will be used. The spread of the local anesthetic will appear hypoechoic on ultrasound. Linear probe will be used.
  For spinal anesthesia levobupivacaine will be placed in the subarachnoid space at lumbar vertebrae 3/4 level using 25 G spinal needle.
  Arms: Extracapsular hip fracture FEMORAL BLOCK; Intracapsular hip fracture FEMORAL BLOCK
Procedure: FIC peripheral nerve block with spinal anesthesia — Suprainguinal approach will be performed. At first, one needs to detect anterior inferior iliac spine, sartorius and internal oblique muscles creating a bow-tie. Deep circumflex iliac artery will be seen between transversus abdominis and iliacus muscle. Then needle needs to be inserted in-plane and 40mL of levobupivacaine 0.25% administered along the fascial plane so that fascia separates from iliacus muscle. The needle is inserted from caudal to cranial, to achieve the widest possible spread of local anesthetic under the fascia, to the cranial side, as this reaches both lateral femoral cutaneous nerve and femoral nerve. The spread of anesthetic will appear hypoechoic on ultrasound. For spinal anesthesia levobupivacaine will be placed in the subarachnoid space at lumbar vertebrae 3/4 level using 25 G spinal needle.
  Arms: Extracapsular hip fracture FASCIA ILIACA BLOCK; Intracapsular hip fracture FASCIA ILIACA BLOCK
Procedure: Fentanyl (IV) with spinal anesthesia — A total dose of 2 mcg/kg of fentanyl will be given to patients before positioning to spinal. For spinal anesthesia levobupivacaine will be placed in the subarachnoid space at lumbar vertebrae 3/4 level using 25 G spinal needle.
  Arms: Extracapsular hip fracture FENTANYL; Intracapsular hip fracture FENTANYL

SUMMARY:
The goal of this clinical trial is to explore the effects of different peripheral nerve blocks in older adults with hip fractures. It will also explore the safety of preoperative administration of peripheral nerve blocks. The main questions this trial aims to answer are:

* which peripheral nerve block is the best regarding analgesia
* which peripheral nerve block eases positioning and decrease time necessary for applying spinal anesthesia?
* which peripheral nerve block is associated with reduced intake of analgesics, both oral and intravenous?
* which peripheral nerve block lasts long enough but does not interfere with the start of physical therapy?
* what medical problems do respondents have during their hospitalization, after administration of peripheral nerve blocks, spinal anesthesia and surgery?
* what medical problems arise as a consequence of their complex medical history? Researchers will compare respondents who receive peripheral nerve blocks to those who do not. Those who do not receive blocks will be given fentanyl preoperatively, which was until recently standard at our institution.

All respondents will, in addition to obligatory intraoperative monitoring,:

* be thoroughly examined by anesthesiologists before surgery
* be closely monitored after surgery, until their hospital discharge.

DETAILED DESCRIPTION:
The aging of the population is a global trend. In the elderly population, hip fractures are among the leading reasons for hospitalization and in most cases require surgical treatment. When we talk about hip fractures, we actually mean fractures of the proximal femur, which are classified according to the AO school as extracapsular (trochanteric region) and intracapsular (femoral neck area). Articular fractures (femoral head area) are very rare and not the subject of this study.

Patients with hip fractures, in addition to their advanced age, have numerous comorbidities. That is why mortality rate is high, up to 36% within a year of surgery, and perioperative care of such patients is a challenge for everyone involved in their treatment, especially surgeons and anesthesiologists. Despite this, to this date our institution has no protocol that would ensure standardization of the care in perioperative period, although this is recommended by professional societies. That is why we designed this study, in which we emphasize use of regional anesthesia in elderly patients.

The goal of this clinical trial is to promote usage of peripheral nerve blocks. Based on our clinical experience, peripheral nerve blocks act as aids for spinal anesthesia positioning and are a crucial part of peri-operative multimodal analgesia protocols in elderly patients scheduled for hip fracture surgery.

We believe that our results will show that peripheral nerve blocks decrease pain and amount of analgesics used in perioperative period, per mouth as well as intravenously. However, in order to include their use into standard operating protocols, we need to determine which block is the best for our group of patients, considering different types of fractures and types of surgeries. We also need to determine which block provides the best analgesia, both for positioning for spinal anesthesia and postoperatively, which block lasts the longest, while not interfering with the start of physical therapy and not prolonging hospital stay.

Primary outcome of this research is to determine pain. It will be determined using visual analogue scale, at rest and dynamically, while leg is being passively raised for 15˚.

Secondary outcomes are: patient reported outcome using EQ-5D-5L, time for the performance of blocks, ease of positioning and time to positioning to spinal, as well as time for the performance of spinal anesthesia, time until the first rescue analgesia and total analgesics used, total duration of blocks, level of motor blockade and time of the initiation of physical therapy, as well as any adverse effects until hospital discharge.

After meeting our inclusion and exclusion criteria, patients will be offered to participate in the research, as respondents. After signing informative consent, they will be randomized into one of four groups, 3 interventional and one control group. Each group will have an equal number of subjects with intracapsular and extracapsular hip fractures. Respondents will not know to which group they have been randomized, nor will the surgeons, nurses and anesthesiology residents. Anesthesiologists will therefore be considered as the study supervisors. Respondents will be closely monitored until hospital discharge.

Anesthesiologist's examination before the surgery will consist of recording body weight and height, determining BMI, noting down history and comorbidities using ASA status, frailty score (Clinical Frailty Test), cognitive status (Mini Mental State Exam), laboratory results (L, WBC, CRP, IL-6, Hb, Htc, ferritin, TSAT, urea, creatinine, eGFR, PLT, PV, INR, APTV, electrolytes) and introducing EQ-5D-5L to respondents. Preoperative fasting will be ensured (6 - 8 hours), clear liquids allowed up to 2 hours before surgery. Upon arrival to the operating block, in the preparation room, respondents will be analgosedated with esketamine 5mg and fentanyl 50 mcg for the administration of peripheral nerve block. Application of peripheral nerve block will be made using ultrasound (linear or curvilinear probe, depending on the block) and regional needles (Pajunk, 21G, length 100 mm). Respondents will be monitored all the time and 20 minutes after administration of the block they will be asked to answer EQ-5D-5L for the second time. After that, they will be positioned for spinal in sitting position. 5 minutes after the spinal they will be asked EQ-5D-5L for the third time and then transported to the operating room. Before the incision, cefazoline and tranexamic acid will be administered. Respondents will be lightly to moderately sedated during surgery (RASS -2 to -3), with propofol and esketamine, sequenced. Normovolemia will be maintained. Intraoperative hypotension will be treated with ephedrine, phenylephrine or norepinephrine. Normothermia will be maintained using passive heating (active if necessary) and body temperature will be measured. Multimodal analgesia will be continued with paracetamol, ketoprofen, dexamethasone and MgSO4. Granisetron will be given as well. Postoperatively, they will answer EQ-5D-5L 4 more times: upon leaving recovery room and operative block, 6 hours after the surgery, 24h and 48h after.

Postoperatively, time until the rescue dose of analgesics will be noted. Analgesics, when necessary, will be introduced in this order: Paracetamol 1 g iv., Diclofenac 75 mg im., Tramadol 50 mg iv., Morphine 2 - 5 mg sc. or iv. After respondents start taking fluids and food per mouth (after 1 hour of receiving fluids, food can be given, or according to the patient's tolerance, but as soon as possible), they can start using analgesics orally. Laboratory results will be done 24h after the surgery, as well as MMSE.

Bromage test for motor blockade will be performed 20 minutes after the block, upon exit from the recovery room, 6h, 24h and 48h after the surgery. Respondents' ability to participate in physical therapy will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

* both sexes
* 60 years old and older
* diagnosed with a hip fracture resulting from low-energy trauma
* scheduled surgery.

Exclusion Criteria:

* polytraumatized patients
* dementia and acute psychosis patients
* patients for whom spinal anesthesia is contraindicated
* patients with severe renal failure
* patients for whom intravenous administration of tranexamic acid is contraindicated
* patients with proven allergy and contraindications to dexamethasone, non-steroidal anti-rheumatic drugs, opioid analgesics, magnesium sulfate.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain relief | 20 minutes after application of the local anesthetic
  The primary outcome measures of this research is pain relief after the administration of peripheral nerve block. Pain will be measured using VAS scale, as a part of one of EQ-5D-5L, at rest and during passive 15˚ leg rising. VAS is the most commonly used scale for pain measurement. VAS ratings (100-mm) of 0 to 4 mm will be considered as no pain; 5 to 44 mm as mild pain; 45 to 74 mm as moderate pain and 75 - 100 mm as severe pain. Cut off values for VAS vary depending on the context and the population. However, 33% decrease in pain is a reasonable standard for determining that a treatment provides meaningful relief.

SECONDARY OUTCOMES:
Health Outcome | before application of the block, 20 minutes after application of the block, 5 minutes after application of spinal anesthesia, 2 hours after the operation (upon leaving the recovery room), 6 hours, 24 hours and 48 hours after the operation.
  Qualitative measure of health outcome will be measured using EQ-5D-5L. Respondents will use it as a self-report, self-complete measure 7 times.
Time for the performance of peripheral nerve block | Before surgery.
  Upon arrival to the block room, respondents need to be monitored, with iv. access obtained, and positioned appropriately. Since these are peripheral nerve blocks, only sterile gloves and antiseptic cleaning solution should be used. A local anesthetic is injected near a specific peripheral nerve, in proximity of a tendon or underneath the fascia. This is achieved using anatomical landmarks and ultrasound guidance. Time for clean up post procedure is also calculated into time to perform blocks. This is measured in minutes.
Time for the performance of spinal anesthesia in a sitting position | Before surgery
  Time to perform spinal anesthesia will be measured in minutes. This interval can be broken down into: monitoring patients, preparing equipment, sitting the patient up, preparing the skin and administering intrathecal injection. This time will be measured in minutes. We will also record ease of positioning respondents to spinal using EOSP score (0 - 3, with higher scores indicating greater ease of positioning and less discomfort), with special emphasis given to time for positioning patients into sitting position (in minutes).
Rescue analgesics | After surgery, up to 48 hours
  We will note the time until patients start asking for analgesics (in minutes) and total quantity of analgetics used (in morphine equivalents).
Duration of peripheral nerve blocks | 20 minutes after the block and 6 hours, 24 hours and 48 hours post surgery
  We will note down total duration of blocks (in hours). We will assess motor blockade using Bromage scale.
Time to the start of physical therapy | After surgery, up to 48 hours
  We will note down when respondents start exercising in bed - passively or actively, sitting - assisted or independently, when they are verticalized - assisted or independently, and when they start walking with aids - assisted or independently.
Development of complications | From the admission, until hospital discharge.
  We will note any adverse effects, if they arise. Complications can be consequences of trauma itself, peripheral nerve blocks, spinal anesthesia and operation itself.
Postoperative nausea | After surgery, up to 48 hours
  Since nausea usually accompanies pain, it will be assessed using VAS scale. 0 is for no nausea and 10 is worst nausea with retching - 20 minutes after application of the block, 5 minutes after application of spinal anesthesia, 2 hours after the operation (upon leaving the recovery room), 6 hours, 24 hours and 48 hours after the operation. Cut off value of 40 will be used as a critical threshold triggering administration of rescue medication.
Anxiety | After surgery, up to 48 hours
  Since anxiety usually accompanies pain, it will be assessed using VAS scale. 0 is for no anxiety and 10 is worst possible anxiety. It will be monitored 20 minutes after application of the block, 5 minutes after application of spinal anesthesia, 2 hours after the operation (upon leaving the recovery room), 6 hours, 24 hours and 48 hours after the operation. Cut off value of 40 will be used as a critical threshold triggering administration of rescue medication.
Quality of recovery | Before and 24 hours after the surgery
  QoR-15 will be introduced to patients the day before, as a measure of baseline status, and 24 hours after the surgery, as a measure of quality of recovery after anesthesia and surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Saric Jadrijev, MD, Principal Investigator — Department of Anaesthesiology and Intensive Care, University Hospital of Split; Ruben Kovac, MD, Study Chair — Department of Anaesthesiology and Intensive Care, University Hospital of Split; Marija Kljucevic, MD, Study Chair — Department of Anaesthesiology and Intensive Care, University Hospital of Split; Petra Bajto, MD, Study Chair — Department of Anaesthesiology and Intensive Care, University Hospital of Split; Meri Mirceta, MD, Study Chair — Department of Anaesthesiology and Intensive Care, University Hospital of Split; Ana Maria Mitar, MD, Study Chair — Department of Anaesthesiology and Intensive Care, University Hospital of Split; Ana Bego, MD, Study Chair — Department of Anaesthesiology and Intensive Care, University Hospital of Split; Josipa Modric, MD, Study Chair — Department of Anaesthesiology and Intensive Care, University Hospital of Split; Nikola Delic, MD, PhD, Study Chair — Department of Anaesthesiology and Intensive Care, University Hospital of Split; Toni Kljakovic-Gaspic, MD, PhD, Study Chair — Department of Anaesthesiology and Intensive Care, University Hospital of Split; Nikola Kljucevic, MD, PhD, Study Chair — Department of Surgery, University Hospital of Split; Boris Luksic, MD, PhD, Study Chair — Department of Surgery, University Hospital of Split
Locations (1):
- University Hospital of Split, Split, Croatia

REFERENCES:
- [Background] Regnault P. The hypoplastic and ptotic breast: a combined operation with prosthetic augmentation. Plast Reconstr Surg. 1966 Jan;37(1):31-7. No abstract available. PMID 5903218
- [Background] Seman AL, Pewen WF, Fresh LF, Martin LN, Murphey-Corb M. The replicative capacity of rhesus macaque peripheral blood mononuclear cells for simian immunodeficiency virus in vitro is predictive of the rate of progression to AIDS in vivo. J Gen Virol. 2000 Oct;81(Pt 10):2441-2449. doi: 10.1099/0022-1317-81-10-2441. PMID 10993932
- [Background] Kim JH, Ju EM, Lee DK, Hwang HJ. Induction of apoptosis by momordin I in promyelocytic leukemia (HL-60) cells. Anticancer Res. 2002 May-Jun;22(3):1885-9. PMID 12168888
- [Background] Nouadje G, Rubie H, Chatelut E, Canal P, Nertz M, Puig P, Couderc F. Child cerebrospinal fluid analysis by capillary electrophoresis and laser-induced fluorescence detection. J Chromatogr A. 1995 Nov 24;717(1-2):293-8. doi: 10.1016/0021-9673(95)00747-3. PMID 8520681
- [Background] Stal P, Hultcrantz R. Iron increases ethanol toxicity in rat liver. J Hepatol. 1993 Jan;17(1):108-15. doi: 10.1016/s0168-8278(05)80530-6. PMID 8445209
- [Background] McCaffrey TV, Olsen KD, Yohanan JM, Lewis JE, Ebersold MJ, Piepgras DG. Factors affecting survival of patients with tumors of the anterior skull base. Laryngoscope. 1994 Aug;104(8 Pt 1):940-5. doi: 10.1288/00005537-199408000-00006. PMID 8052078